CLINICAL TRIAL: NCT06367283
Title: Metformin Treatment of Patients with Hand Osteoarthritis: a Randomised, Placebo-controlled Trial
Brief Title: Metformin Treatment of Patients with Hand Osteoarthritis
Acronym: METRO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Marius Henriksen (Other)
Responsible Party: Sponsor-Investigator, Marius Henriksen, Professor, Frederiksberg University Hospital
Organization: Frederiksberg University Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2023-509181-38-00
Record Dates: First submitted 2024-04-03; First posted 2024-04-16 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Hand Osteoarthritis
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Metformin (Experimental)
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Metformin — Metformin will be initiated at 500 mg once daily with breakfast meal. The dose will be increased with 500 mg every week until 2 g/day is reached, distributed as 1000 mg every morning and evening, together with a meal. If the subject cannot tolerate the maximum dose (2 g/day), the maximal tolerated dose will be given. The treatment period including titration is 16 weeks.
  Arms: Metformin
Drug: Placebo — Participants in the placebo group will receive a placebo tablet identical to the metformin tablet
  Arms: Placebo

SUMMARY:
To compare metformin (2 g daily), or maximum tolerated dose, for 16 weeks with placebo as a treatment of hand osteoarthritis symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years
2. Hand OA according to the ACR criteria
3. Average finger (2 to 5) pain ≥4 on a 0-10 numeric rating scale (NRS where 10 is worst pain) over the past 30 days
4. Metformin naive

Exclusion Criteria:

Comorbidities

1. History of, or current signs of medical disease that may affect joints, e.g. rheumatoid arthritis, gout, psoriatic arthritis
2. Psoriasis
3. Known malignancy (except successfully treated squamous or basal cell skin carcinoma)
4. Drug or alcohol abuse in the last year
5. Existing nerve entrapment syndromes (e.g. carpal tunnel syndrome)
6. Known diabetes
7. Generalised pain syndromes such as fibromyalgia
8. Known peripheral neuropathies
9. Known allergies towards the interventions
10. Gastric bypass or other malabsorption syndrome
11. In case of pharmacological weight loss medication (e.g. glucagon like peptide-1 (GLP-1) analogues) or pharmacological osteoporosis medication, dosage must have been stable for 3 months without any plan of up-titration during the study period
12. Any other condition or impairment that, in the opinion of the investigator, makes a potential participant unsuitable for participation or obstructs participation e.g. psychiatric disorders.

    Surgical history
13. History of hand surgery in the target hand within 12 months prior to enrolment
14. History of arthroplasty, arthrodesis or surgical treatment of thumb base osteoarthritis in the target hand

    Management strategies
15. Use of systemic corticosteroids equivalent of ≥ 7.5 mg prednisolone daily within 3 months
16. Treatment with denosumab (Prolia/Xgeva)
17. Participation in experimental device or experimental drug study 3 months prior to enrolment
18. Intra-articular treatments of any kind of any joint of the target hand 3 months before inclusion
19. Current use of synthetic or non-synthetic opioids
20. Planning to start other treatment for hand OA in the study participation period
21. Planned CT scan with iodine contrast
22. Scheduled surgery on upper extremity of the target hand during study participation
23. Scheduled surgery requiring pause of metformin, e.g. surgery in general anaesthesia, during study participation

    Reproductive system
24. Pregnancy
25. Planned pregnancy within the study period, 3 months after end of study treatment for female fertile participant and 6 months after end of study treatment for male participant
26. Insufficient anti-conception therapy for female fertile participants within the study period and 3 months after end of study treatment

    * Sufficient anti-conception therapy consists of intra-uterine device (coil), hormonal anti-conception (birth control pills, implant, intra-uterine system, dermal patch, vaginal ring, or injections) or sexual abstinence
    * Female participants are considered infertile if they are postmenopausal or if they have undergone surgical sterilisation (bilateral salpingectomy, hysterectomy or bilateral oophorectomy)
    * Postmenopausal state is defined as no menses for 12 months without alternative medical cause before inclusion in the study
27. Insufficient anti-conception therapy for male participants within the study period and 6 months after end of study treatment

    * Sufficient anti-conception therapy consists of condom or sexual abstinence
    * Male participants are considered sterile if they have undergone surgical sterilisation (vasectomy)
28. Breast-feeding

    Blood analysis
29. Positive anti-cyclic citrullinated peptide (>10 kU/L)
30. eGFR <60 ml/min/1.73 m2
31. Vitamin B12 deficiency < 200 pmol/L
32. Hba1c ≥ 48 mmol/mol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Finger pain | Week 16
  Change from baseline in Visual Analogue Scale (VAS) finger joint pain of the target hand after 16 weeks of treatment

SECONDARY OUTCOMES:
Function | Week 16
  Change from baseline after 16 weeks of treatment in physical function assessed by Australian/Canadian Osteoarthritis Hand Index (AUSCAN) physical function subscale
Thumb base pain | Week 16
  Change from baseline after 16 weeks of treatment in Visual Analogue Scale thumb base pain of the target hand
Hand pain | Week 16
  Change from baseline after 16 weeks of treatment in pain of both hands assessed by Australian/Canadian Osteoarthritis Hand Index hand pain subscale
Physician tender joint count | Week 16
  Change from baseline after 16 weeks of treatment in joint activity of the target hand assessed by physician tender joint count
Patient global assessment | Week 16
  Change from baseline after 16 weeks of treatment in Visual Analogue Scale patient global assessment
Quality of life assessed by the European Quality of life - 5 dimensions (EQ-5D) scale | Week 16
  Change from baseline after 16 weeks of treatment in quality of life assessed by the European Quality of life - 5 dimensions scale
Hand strength | Week 16
  Change from baseline after 16 weeks of treatment in hand strength of the target hand assessed by a grip dynamometer
Number of treatment responders | Week 16
  Responders will be identified according to OMERACT-OARSI criteria, defined as (1) improvement in finger pain (primary outcome) or function (secondary outcome) ≥50% and an absolute change ≥20 mm; or (2) improvement of ≥20% with an absolute change ≥10 mm in at least two of the following three: finger pain (primary outcome), function (secondary outcome), and patient global assessment (secondary outcome).

OTHER OUTCOMES:
Stiffness of both hands | Week 16
  Change in stiffness of both hands measured on the Australian/Canadian Osteoarthritis Hand Index (AUSCAN) stiffness subscale
Composite of pain, function and stiffness | Week 16
  Change in pain, function and stiffness of both hands measured composite on the Australian/Canadian Osteoarthritis Hand Index (AUSCAN) Hand Index Score
Physical function | Week 16
  Change in physical function of both hands assessed by the Health Assessment Questionnaire Disability Index (HAQ-DI)
Physician global assessment | Week 16
  Change in physician global assessment of disease activity of hand OA in the target hand measured on a Visual Analogue Scale (VAS) scale
Swollen joint count | Week 16
  Change in physician swollen joint count of the target hand
Fatigue | Week 16
  Change in fatigue measured on a Visual Analogue Scale (VAS) scale
Sleep quality | Week 16
  Change in sleep quality measured on the Pittsburgh Sleep Quality Index (PSQI)
Absence or presence of inflammation of target hand | Week 16
  Change in absence or presence of inflammation of the target hand as measured by ultrasound (US)
Change in use of analgesics | Week 16
  Change in use of analgesics measured as the use of paracetamol and NSAIDS
Inflammatory biomarker | Week 16
  Change in hsCRP mg/L
Metabolic outcomes | Week 16
  Change in HbA1c mmol/mol
Metabolic outcomes | Week 16
  Change in lipids mmol/L
Vitamin K | Week 16
  Change in vitamin K and dephospho-uncarboxylated matrix Gla-protein ((dp)ucMGP) pmol/L
Proteomics | Week 16
  Change in mass-spectrometry based proteomics

CONTACTS AND LOCATIONS:
Locations (1):
- The Parker Institute, Bispebjerg and Frederiksberg hospital, Copenhagen, Frederiksberg, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Data sharing plan Individual participant data that underlie the results reported in this study and analytic code will be availa-ble from Henning Bliddal (henning.bliddal@regionh.dk) once all planned analyses have been completed and published. The request will be considered on individual basis. Consent for data sharing was not obtained, but the dataset is anonymised, and risk of reidentification is very low. The study protocol and statistical analysis plan are part of the manuscript. The informed consent form is available upon re-quest.

REFERENCES:
- [Derived] Madsen KS, Henriksen M, Dossing A, Poulsen AS, Oscar R, Kragstrup T, Ellegaard K, Knop FK, Boesen M, Hunter DJ, Christensen R, Bliddal H. Metformin treatment for patients with hand osteoarthritis: protocol for the multicentre, randomised, placebo-controlled METRO trial. BMJ Open. 2025 Mar 26;15(3):e093831. doi: 10.1136/bmjopen-2024-093831. PMID 40139705